CLINICAL TRIAL: NCT00779350
Title: A Study to Compare the Relative Bioavailability of Ranbaxy and Pfizer Formulations of Sertraline 100 mg Tablets in Healthy Adult Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Sertraline Hydrochloride 100mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10540323
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence sertraline 100 mg tablets fasting conditions
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sertraline 100 mg tablets of ranbaxy
  Interventions: Drug: sertraline 100 mg tablets
- 2 (Active Comparator): Zoloft® 100 mg tablets
  Interventions: Drug: sertraline 100 mg tablets

INTERVENTIONS:
Drug: sertraline 100 mg tablets

SUMMARY:
The purpose of this study was to evaluate the relative bioavailability of the test formulation of sertraline 100 mg tablets with an already marketed reference formulation Zoloft® 100 mg tablets (Pfizer), under fasted conditions in healthy male and female adult subjects.

DETAILED DESCRIPTION:
This randomized, single-dose, two-way, crossover study was conducted to compare the relative bioavailability of two formulations of 100 mg sertraline hydrochloride tablets under fasting conditions. The study was conducted with 36 (30 completing) healthy adults in accordance with protocol No.

10540323(Revision 0). In each study period, a single 100 mg dose was administered to the subjects following an overnight fast of at least 10 hours. The test formulation was Ranbaxy Research Laboratories's Sertraline Hydrochloride 100 mg Tablets and the reference formulation was ZOLOFT® (sertraline hydrochloride) 100 mg Tablets Manufactured by Roerig (Division of Pfizer). The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. There was a 14-day interval between treatments.

Blood samples were collected pre-dose and at intervals over 144 hours after each dose. The plasma samples for all subjects completing both periods of the study were sent to Helen Fassoulas, B.Sc., Director of Operations, Warnex Bioanalytical Services Inc., 3885 boul Industriel, Laval, Quebec, H7LAS3 Canada, Telephone: 450-663-6724, ext. 438, FAX: 450-975-8111 for determination of sertraline plasma concentration.

Statistical analysis was performed by Yetta I. Wilbur, Biostatistician, Novum Pharmaceutical Research Services, 5900 Penn Avenue, Pittsburgh, PA 15206, USA, Telephone: 412-363-3300, Fax: 412-362-5783 to evaluate the relative bioavailability of the test formulation to that of the reference product.

A total of 36 healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-65 years of age (inclusive).
* A body mass index (BMI) of 18-30 kg/m2 inclusive as measured and calculated according to Novum Standard Operating Procedures.
* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
* Signed and dated informed consent form, which meets all criteria of current FDA regulations.
* Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable method of contraception (e.g. condom with spermicide, IUD, hormonal contraceptives) for at least 30 days prior to dosing and during the duration of the study.

Exclusion Criteria:

* If female, pregnant, lactating or likely to become pregnant during the study.
* History of allergy or sensitivity to sertraline hydrochloride or other selective serotonin reuptake inhibitor's (SSRI's), or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction.
* Presence of gastrointestinal disease or history of malabsorption within the last year.
* History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
* Use within 14 days of dosing, or anticipated use during the study, or for 14 days after the last dose of sertraline any monoamine oxidase inhibitors (MAOIs).
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 ml or more) with/n 30 days or plasma within 14 days prior to dosing.
* Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Positive serum pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-08; Primary Completion 2005-08 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html